CLINICAL TRIAL: NCT06837766
Title: Observational Study About Hepatic Toxins Kinetic and Evaluation of Organ Damage in Acute on Chronic Liver Failure (ACLF) Patients: Multicenter Prospective Observational Spontaneous Study
Brief Title: Study About Hepatic Toxins Kinetic and Evaluation of Organ Damage in Acute on Chronic Liver Failure (ACLF) Patients
Acronym: BILIVER2020
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: BILIVER2020; WFR RC 2773286 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-11-28; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-10

CONDITIONS: Acute on Chronic Liver Failure (ACLF)
Keywords: Acute on Chronic Liver Failure (ACLF),; Model for End stage Liver Disease (MELD); Chronic LIver Failure - Consortium Organ Failure (CLIF-C OF); Renal Replacement Therapy (RRT)
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Spontaneous Observational Prospective Multicenter study of all patients admitted to Intensive Care with a diagnosis of Acute on Chronic Liver Failure (ACLF) of grade ≥ 2 for which the use of the system will be authorized extracorporeal purification with DM CYTOSORB. The hypothesis underlying the study is to evaluate whether the modulation of bilirubin and other toxic molecules and mediators, obtainable through the use of systems extracorporeal purification (specifically DM CYTOSORB), may have an impacton the degree of organ failure in patients with ACLF.

The study proposes the compilation of a structured and shared data collection with other Italian Intensive Care Centers which include patients suffering from ACLF (multicenter study) of clinical and laboratory parameters, which are part of normal clinical practice.

DETAILED DESCRIPTION:
The Acute on Chronic Liver Failure (ACLF) according to the definition of the "European Association for the Study of the Liver - Chronic Liver Failure (EASL-CLIF)" formulated in 2014 and derived from the CANONIC study, occurs in patients liver disease with or without a previous history of decompensation, which develops an acute deterioration of pre-existing liver disease (chronic liver disease, compensated or non-compensated cirrhosis). Such deterioration, dependent on one or more acute events, characteristically correlates with non-organ failure only hepatic, but also extrahepatic, and to a high 28-day mortality (>15%). Given the recent definition of ACLF and the ongoing studies on the clinical course, on prognosis and hospital management of these patients, no conclusions yet exist guidelines with high levels of evidence, but only consensus of opinions, formulated mainly from clinical experience or derived from the treatment of cirrhosis or acute liver failure. In the knowledge that the ACLF is one delicate syndrome, over time the importance of an approach has been underlined multidisciplinary team of intensivists, hepatologists, nephrologists, infectious disease specialists and surgeons specialized in transplants. Considering that these patients present with an o more organ failure, the most suitable environment for hospitalization, in particular of those who have high-grade ACLF, it is intensive therapy, which allows support vital functions invasively and carefully monitor him clinical development.

In liver failure the liver loses its physiological ability to purify the blood from endogenous waste substances (ammonium, proinflammatory cytokines, endogenous benzodiazepines and aromatic amino acids), but also its activity biosynthetic and homeostatic; at the moment, however, there is no real one treatment of liver failure, if not transplantation. In fact the only treatment the solution for ACLF is orthotopic liver transplant (OLT); the procedure remains however applicable in a limited number of cases, considering the scarcity of organs available and the frequent presence of contraindications, which prevent the inclusion of these patients on the list.

Therefore, various extracorporeal systems have been developed and tested liver support, which are intended to support liver function and limit/slow down multiple organ failure. The systems developed so far do differ due to the use of different filtration membranes: on the one hand the MARS (Molecular Adsorbent Recirculating System), which, with a technique similar to dialysis, combines kidney support with albumin dialysis through a filter highly selective; on the other, a high-volume plasmapheresis technique with much less selective plasma separation and filtration (Prometheus).

CYTOSORB has been added to these purification systems that work on plasma works on whole blood. Cytosorb is a disposable adsorbent resin cartridge capable of adsorbing an excessive level of cytokines as the blood passes through the device. The use of Cytosorb in patients with ACLF finds its place rational in the fact that it is able to adsorb the excess of cytokines circulating from the blood of patients with severe sepsis, septic shock, multi-organ damage and "systemic inflammatory response syndrome" (SIRS), which is the mechanism supposed to also be the basis of ACLF, it can increase the effectiveness of the therapy standards of support for these patients and improve their prognosis. To this effect the main one is associated with that resulting from the adsorption of excessive levels of myoglobin, free hemoglobin and bilirubin to prevent organ damage and improve the prognosis of patients.

At the moment the role of these systems in the management of ACLF is very limited and the studies carried out have shown mixed results; it is definitely described a improvement of laboratory data (decrease in bilirubin, bile acids, urea, ammonium and creatinine) associated with clinical improvement encephalopathy and hemodynamics, but an increase in survival associated with the use of these systems. It should be noted, however, that these devices were studied in a population with ill-defined ACLF and which therefore would require trials carried out on larger cohorts. It is therefore necessary to study these systems in more depth, than on paper represent a therapeutic possibility and an effective bridge for patients serious patients waiting for a transplant, but, for now, they have not demonstrated effectiveness clinically significant.

The hypothesis underlying the study is to evaluate whether the modulation of bilirubin and other toxic molecules and mediators, obtainable through the use of extracorporeal purification systems (specifically DM CYTOSORB), can affect the degree of organ failure in patients with ACLF; to this end the device in question used by the Doctor on the basis of his clinical judgment in context of daily clinical practice and in a decision-independent manner to include the patient in the study must be authorized by the Management Healthcare. The study proposes the compilation of a structured data collection and shared with other Italian intensive care centers to which affected patients belong from ACLF (multicenter study) of clinical and laboratory parameters, which fall in normal clinical practice.

The primary objective of the study is to evaluate the trend of the main toxins involved in liver failure (bilirubin, bile acids and ammonium) in patients suffering from ACLF.

The secondary objectives of the study are:

1. Observation of the following clinical outcomes:

   I. Liver function: liver enzymes; lactates; coagulation parameters; MELD score e CLIF-OF score. II. Inflammatory state: PCR; PCT; leukocytes. III. Neurological function: degree of encephalopathy. IV. Renal function: urinary output; serum creatinine. V. Cardiovascular function: MAP; need for vasopressors; THERE
2. Incidence of clinical complications and adverse events;
3. Length of stay in Intensive Care Unit;
4. Need for liver transplantation;
5. Survival at 28 days. This study is of a Spontaneous Prospective Observational type, not interventional, multicentre, and will be conducted on all patients admitted to therapy Intensive care with ACLF diagnosis defined according to the criteria established by the study CANONIC of EASL-CLIF1: syndrome, which occurs in patients who already have a chronic liver disease with or without cirrhosis, characterized by acute deterioration of pre-existing liver disease resulting in liver failure and o more extrahepatic organ failure and associated with high mortality at 28 days from onset.

The degree of organ failure is assessed through a score (CLIF-OF-SOFA) born as an adaptation of the SOFA score in a hepatological environment and then simplified in the CLIF-C-OF score.

All patients admitted to the Intensive Care Unit of each year will be enrolled in the study participating center, with a diagnosis of ACLF defined according to the criteria established by the CANONIC study of EASL-CLIF1 that meet the inclusion criteria.

The study is observational, non-interventional and provides for each patient including a collection of demographic, clinical and laboratory parameters that fall within normal clinical practice (see CRF). This data collection will concern all patients suffering from ACLF grade ≥ 2 and undergoing haemoabsorptive treatment with Cytosorb as required by clinical practice in accordance with the judgment of Doctor and the information reported in the Technical Data Sheet of the aforementioned device (DM Cytosorb).

Cytosorb being proposed in addition to the standard therapy it includes early identification and treatment of the precipitating event (trigger) if identified , supportive therapy to ensure haemodynamic stabilisation , therapy for the treatment of insufficiency renal, it is underlined that the above-listed concomitant therapies are permitted by protocol and are part of normal clinical practice. In particular, in the case of concomitant renal failure , the cartridge Cytosorb can be inserted in series on the "Continuous" dialysis circuit Renal Replacement Therapy" (CRRT). Also as required by the Commission Company devices, the use of Cytosorb requires compilation by the doctors of a follow-up card (Cytosorb_follow-up card) for each patient treated which specifies the duration of the treatment, number of cartridges used, days of hospitalization in the ICU, days of total hospitalization and outcome (transfer to another department or death).

The personnel designated by the Investigator must report the requested information from the protocol on the Data Collection Form (CRF). The CRF data will be entered into a database by personnel designated by the experimenter. At the end of the data entry, the control and the data validation.

The characteristics of the patients enrolled in the study will be reported in tables synthesis.

Descriptive statistical analyzes will be used to describe the data collected: le continuous variables will be described by means, standard deviation (or median and interquartile distance), minimum values, maximum values and percentiles; discrete variables or nominal frequencies will be described and summarized using absolute frequencies and frequencies relative percentages. The parameters analyzed will be bilirubin, bile acids and ammonium, liver enzymes, lactates and coagulation parameters; MELD score and CLIF-OF score; PCR, PCT, leukocytes; degree of encephalopathy; urinary output, serum creatinine; MAP, need for vasopressors and IC.

At the various visits, the values regarding clinical parameters and tests will be recorded laboratory and blood gas analyzes in order to quantify the extent of the variations through absolute values and relative percentage deviations compared to the baseline value.

a) the incidence will be calculated, with relative confidence intervals (95% CI), of clinical complications and adverse events, b) length of stay in Intensive Care, c) need for liver transplantation. Survival at 28 days will be estimated using Kaplan Meier curves. Data will be analyzed using IBM SPSS Chicago-Illinois statistical software (ver. 22.0).

Prospective observational study that aims to evaluate whether the modulation of bilirubin and other toxic molecules and mediators, obtainable through the use of extracorporeal purification systems (specifically DM CYTOSORB), can affect the degree of organ failure in patients with ACLF. A preliminary evaluation of the case series concerning patients affected by ACLF relating to the Italian intensive care centers participating in the study allows for hypothesize that, within 48 months of the start of the program, they can be recruited and followed approximately 40 patients with the inclusion characteristics indicated in paragraph 3.2.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute hepatic decompensation on chronic liver disease with grade ACLF ≥ 2 (diagnosable in the presence of at least two defined organ failures according to the CLIF-C-OF score);
* hemoabsorbent treatment with Cytosorb;
* patients aged ≥ 18 years at the time of diagnosis;
* Informed Consent.

Exclusion Criteria

* patients aged < 18 years;
* fulminant liver failure;
* chronic end-stage liver failure with chronic encephalopathy and/or chronic refractory ascites;
* acute on chronic hepatic decompensation with grade 0 or 1 ACLF;
* clinical signs or history of congestive heart failure (NYHA class 3-4 before the acute phase of the disease or documented EF < 35% or PCWP > 18 mmHg) or acute coronary syndrome
* state of immunosuppression (rheumatological and immunological diseases, HIV, immunosuppressive therapy);
* previous organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Intensive Care Unit of each year will be enrolled in the study participating center, with a diagnosis of ACLF defined according to the criteria established by the CANONIC study of EASL-CLIF1 that meet the inclusion criteria listed before.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | Baseline, day 1, day 2, day 3, day 7, day 8, until completion of the study (average 10 days).
  The hypothesis underlying the study is to evaluate whether the modulation of bilirubin and other molecules (bile acids and ammonium) and toxic mediators (citokynes), obtainable through the use of extracorporeal purification systems with DM CYTOSORB, can affect the degree of organ failure in affected patients from ACLF.

SECONDARY OUTCOMES:
Secondary outcome | From admission to intensive care up to 28 days.
  Incidence of clinical complications and adverse events.
Third otucome | From admission to intensive care up to 28 days.
  Length of stay in Intensive Care Unit.
Fourth outcome | From admission to intensive care up to 28 days.
  Need for liver transplantation.
Fifth outcome | From admission to intensive care up to 28 days.
  Survival at 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Siniscalchi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - Azienda Ospedaliero-Universitaria Ospedale Riuniti Umberto I - GM Lancisi - G Salesi, Ancona, Ancona, Ancona
  - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna, Bologna
  - Anestesia e Rianimazione 2, Ospedale Niguarda Ca' Granda, Milano, Milan, Milano